CLINICAL TRIAL: NCT03005080
Title: The Utility of Pharmacogenetic Testing in Managing Children With Persistent Gastroesophageal Reflux Disease Despite Therapy
Brief Title: Pharmacogenetic Testing in Children With Persistent Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Imad Absah, Imad Absah, M.D., Mayo Clinic
Other Study IDs: 16-007265
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will use a 22 gene pharmacogenomics panel on 30 children with persistent Gastroesophageal Reflux Disease (GERD) who have not responded to therapy.

DETAILED DESCRIPTION:
This study will assess the clinical utility of pharmacogenomics testing in the clinical management of children with refractory GERD, despite adequate therapy and the role of pharmacogenomics in selecting the right acid suppressive therapy based on each patient's symptoms and pharmacogenomics results.

ELIGIBILITY:
Inclusion Criteria:

* persistent gastrointestinal symptoms (GI) suggestive of gastro esophageal reflux disease (GERD) despite adequate therapy
* persistent evidence of abnormal reflux indices' and acid exposure on esophageal multichannel pH impedance study despite adequate therapy
* persistent endoscopic evidence of reflux esophageal disease despite adequate therapy

Exclusion Criteria:

* children with eosinophilic esophagitis diagnosis
* children with any esophageal surgical intervention like fundoplication, tracheoespahgeal fistula repair or esophageal atresia repair
* children with other diseases that can affect the esophagus, like Crohn's disease or food protein-induced enterocolitis syndrome (F-PIES)
* Children who do not have research authorization in their chart

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children <18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects who change medication due to pharmacogenomic results | 12 weeks
Number of subjects who have a repeat scope | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials